CLINICAL TRIAL: NCT01369394
Title: Developing a Computer-based Intervention That Provides Individually-tailored Educational Information for MMR Vaccine-hesitant Parents
Brief Title: Making Decisions About the Measles-Mumps-Rubella Vaccine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Amanda Dempsey, Associate Professor of Pediatrics, University of Colorado, Denver
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 186564
Record Dates: First submitted 2011-06-07; First posted 2011-06-08 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Measles; Mumps; Rubella; MMR Vaccination
Keywords: Measles; Mumps; Rubella; MMR; Prevention; Tailoring; Persuasive communication; Children
MeSH Terms: conditions — Measles; Mumps; Rubella

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tailored information (Experimental): Individuals assigned to the experimental group will receive individually-tailored educational messages.
  Interventions: Other: Behavioral: Computer-based tailoring system
- Untailored information (Active Comparator): Individuals assigned to the control group will receive generic, untailored educational messages.
  Interventions: Other: Behavioral: Computer-based tailoring system

INTERVENTIONS:
Other: Behavioral: Computer-based tailoring system — Both the intervention and control groups will use a computer-based tailoring system to respond to survey questions. The computer-based tailoring system will generate educational messages based on participants' responses to survey questions. The intervention group will receive tailored educational messages, whereas the control group will receive generic educational messages. The tailored and generic educational messages will be presented as to look like web pages. However, the messages will only exist on the study computer, and will not be linked to any "live" server or website.

SUMMARY:
The goal of this study is to determine whether a computer-based intervention that delivers individually-tailored educational messages about the MMR vaccine increases MMR vaccine-hesitant parents' intentions to have their children vaccinated.

DETAILED DESCRIPTION:
This will be a randomized controlled intervention trial for MMR vaccine-hesitant parents of children ages six years and younger who have not yet received the MMR vaccine. Parents will complete a three-item measure that assesses their baseline intentions for having their children vaccinated with MMR. Participants will then fill out a short, computer-based survey that assesses demographic factors, prior experience with MMR, and views about a variety of potential barriers to MMR vaccination. Following the survey, the intervention group (40 parents) will view a series of tailored educational messages resembling web pages that uses their survey data to address at an individual level their specific concerns about the MMR vaccine. The control group (40 parents) will view a series of generic educational messages resembling web pages that is similar in appearance to the intervention, but contains only untailored information about the vaccine. After navigating through these educational messages, MMR vaccination intention will be reassessed using the same three-item measure as for the baseline assessment of vaccination intention. The vaccine administration records of the children of these parents will be accessed after parents' participation in the study to assess whether the MMR vaccine was provided to the child.

ELIGIBILITY:
Inclusion Criteria:

* Parent is greater than or equal to 18 years of age
* Parent has a child 6 years of age or younger
* When asked to describe how he/she feels about getting child vaccinated against MMR, parent responds "I don't want to get my child vaccinated" or "I'm unsure if I want my child to get vaccinated"

Exclusion Criteria:

* Cannot read/speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Parent's intention to vaccinate child against MMR | Date of intervention (one day)
  Parent will rate his/her intention to have child vaccinated against MMR using a Likert scale before and after the intervention.

SECONDARY OUTCOMES:
Use of the intervention | At the time of intervention participation
  We will assess the number of pages viewed and time spend per page for each participant viewing the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Dempsey, MD, PhD, MPH, Principal Investigator — Children's Outcomes Research Program
Locations (1):
- UMHS Outpatient Pediatrics, Ann Arbor, Michigan, United States